CLINICAL TRIAL: NCT04370093
Title: Pathogenesis of Uric Acid Nephrolithiasis: Role of Pioglitazone/Weight Loss
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Khashayar Sakhaee, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STU-2019-0907
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Nephrolithiasis, Uric Acid
Keywords: Biomedical Sciences
MeSH Terms: conditions — Nephrolithiasis | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Pioglitazone Drug (including Placebo) (Experimental): 45 mg/day- one pioglitazone tablet once daily throughout the 24 weeks of the study
  Interventions: Drug: Pioglitazone 45 mg
- Weight Loss, Behavioral (Experimental): Weight loss following the Group Lifestyle Balance Program based on the Diabetes Prevention Program that utilizes cognitive behavioral strategies (goal setting, problem solving, self-monitoring, stimulus control),and provides written education materials to support health and nutrition behavior changes for weight management and disease prevention.
  Interventions: Behavioral: Weight Loss
- Pioglitazone + Weight Loss (Other): Pioglitazone 45 mg/day + Weight Loss following the Group Lifestyle Balance Program based on the Diabetes Prevention Program that utilizes cognitive behavioral strategies (goal setting, problem solving, self-monitoring, stimulus control),and provides written education materials to support health and nutrition behavior changes for weight management and disease prevention.
  Interventions: Other: Pioglitazone + Weight Loss

INTERVENTIONS:
Drug: Pioglitazone 45 mg — 45 mg/day- one pioglitazone tablet once daily throughout the 24 weeks of the study
  Arms: Pioglitazone Drug (including Placebo)
Behavioral: Weight Loss — Weight loss following the Group Lifestyle Balance Program based on the Diabetes Prevention Program that utilizes cognitive behavioral strategies (goal setting, problem solving, self-monitoring, stimulus control),and provides written education materials to support health and nutrition behavior changes for weight management and disease prevention.
  Arms: Weight Loss, Behavioral
Other: Pioglitazone + Weight Loss — Pioglitazone + Weight loss following the Group Lifestyle Balance Program based on the Diabetes Prevention Program that utilizes cognitive behavioral strategies (goal setting, problem solving, self-monitoring, stimulus control),and provides written education materials to support health and nutrition behavior changes for weight management and disease prevention.
  Arms: Pioglitazone + Weight Loss

SUMMARY:
The investigators will randomize overweight and obese iuan patients to Pio (45 mg/day, highest approved dose or placebo), WL (10% of body weight, following the established program used in the Diabetes Prevention Program), or Pio+WL. Participants will be evaluated at baseline and after 24 weeks of intervention while on a fixed metabolic diet to exclude the confounding effects of diet and perspiration. The primary endpoint will be change in upH, and multiple additional endpoints (serum, urine, imaging) will be assessed.

DETAILED DESCRIPTION:
In IUAN patients, the investigator will compare 1. PPAR activation; 2. weight loss; or 3. combination; on urine acid-base parameters relevant to UA stone risk. The investigator will assess the effect of these interventions on fat distribution, insulin sensitivity, and serum adiponectin, and correlate these changes with urine chemistry.

Hypothesis: Weight loss + TZD independently result in durable changes in urine chemistry.

Significance: Epidemiology of uric acid nephrolithiasis: Nephrolithiasis is an increasingly prevalent condition that leads to significant pain1, work productivity loss2, reduced quality of life3, urinary tract infection4, chronic kidney disease5,6 and end-stage renal disease7. In the U.S., nephrolithiasis prevalence doubled in the past 30 years to a level similar to diabetes, and is the most expensive non-malignant urologic condition (2006 U.S. annual cost: $10 billion)8. Compared with other stone types, uric acid stones recur at a higher rate9, lead to more CKD10, and comprise a rising fraction of stones11,12 , in part due to the growing prevalence of obesity and diabetes13-18. The single most important pathogenic factor in human IUAN is an overly acidic urine, promoting protonation of urate to the insoluble UA16,19. In previously completed NIH-supported studies, the Investigator identified increased net acid excretion and blunted ammoniagenesis to be the principal metabolic defects underlying aciduria in humans IUAN and in rodent models of IUAN risk16,18,20-23. Treatment has been empirical urinary alkalinization24 which is efficacious but has not changed since 1986. Limitations include frequent dosing25, need for high dose in obese patients26, medication intolerance27, and need for periodic urine collections disliked by patients. Therapy that targets the underlying pathophysiologic defect rather than urinary chemistry is directly needed. The Investigator showed that the thiazolidinedione (TZD) pioglitazone that activates PPAR, improves systemic and urinary abnormalities in IUAN including impaired excessive acid excretion and ammoniagenesis, and results in a rise in UpH. TZD treatment of rodent IUAN model shows similar improvements28. The Investigator may have a therapy targeting the underlying pathobiology.

The translational potential of our regimen is extremely high and immediate. If combined TZD and weight loss (Aim) are efficacious in reducing stone risk, one can move straight to a clinical trial using hard outcomes such as stone events, and stone count by imaging to test this regimen. None of these maneuvers requires FDA approval to initiate. Patients will then have instant control of urinary chemistry with empiric alkali therapy (existing therapy), but also a chance to achieve more lasting improvement with TZD and weight loss, which reverses the pathophysiology. Separately, adiponectin (APN) receptor agonists are being developed as potential pharmacological agents for the management of metabolic syndrome complications including diabetes and dyslipidemia29,30. If approved, such agents could be tested as therapy for aciduria in the metabolic syndrome if adiponectin mediates the impact of TZD on renal ammoniagenesis.

UA nephrolithiasis is the clinically palpable sentinel of some complex underlying systemic pathophysiology; hence the impact of these studies extends beyond UA stones. The Investigator is examining a novel multi-organ paradigm of increased acid production from the gut that escapes hepatic metabolism, and ending up as an acid load imposed on the kidney. When compounded with renal ammoniagenesis defect, this leads to aciduria and UA lithogenesis. The Investigator will address some fundamental pathobiologic mechanisms of the metabolic syndrome. Due to the time and budget limits, the Investigator will concentrate our efforts to yield informative data; hence the renal focus. Our long-term goal is to use this as a portal to study multiple aspects of the gut, hepatic, and adipose pathophysiology of the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

Idiopathic uric acid nephrolithiasis, with last stone analysis showing that stone has >90% uric acid in composition Age >21 years Any gender, race/ethnicity (from weight loss), but weight <165 Kg (to fit into MR instrument); eGFR>60ml/min/1.73 m2

Exclusion Criteria:

Bariatric surgery, chronic diarrhea, recurrent UTIs current insulin use use of a thiazolidinedione in past 2 years contraindication to thiazolidinedione use (liver dz, pedal edema, CHF NYHA class III/IV, no contraception) Bladder cancer Use of SGLT2-i, GLP-1 analogs, gemfibrozil, topiramate, rifampin Hba1c > 8.5%

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Urine pH | 24 weeks
  24-hour urine pH is the main determinant of uric acid stone formation and recurrence.

SECONDARY OUTCOMES:
Urine Ammonium/Net Acid Excretion | 24 weeks
  The ratio of urine ammonium to net acid excretion (NH4+/NAE) is a key pathophysiologic risk factor to uric acid stone formation. This is calculated from 24 hr urine ammonium and 24 hr urine net acid excretion.
Urine Net Acid Excretion/Sulphate | 24 weeks
  Urine Net Acid Excretion to Sulphate ratio represents the diet-independent fraction of acid excreted. This is calculated from 24 hr urine net acid excretion and 24 hr urine sulphate.
Supersaturation Index of Uric Acid | 24 weeks
  Supersaturation Index of Uric Acid is a calculated parameters that indicates the degree of urinary saturation with respect to uric acid.

CONTACTS AND LOCATIONS:
Overall Officials: Khashayar Sakhaee, MD, Principal Investigator — UTSW
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States